CLINICAL TRIAL: NCT04924842
Title: Epidemiology of CoV-2 SARS Infections: Dynamics of Community Contamination in Children and Adults - Impact of Variants
Brief Title: COVID-19 - SARS-CoV-2 Community Contamination in Children and Adults - Impact of Variants (Dyn3CEA - Nosocor Phase 2)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0564
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Infection Viral
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Hospitalized children, 0 to 17 years of age, 30 subjects, consecutive sample survey, recruitment in quotas of five age ranges.
  Interventions: Other: Review of medical file
- Adults: Hospitalized adults, 18 years and above, 60 matched subjects
  Interventions: Other: Phone call interview

INTERVENTIONS:
Other: Review of medical file — Review of medical patient file, including patient tracing, brief summary of the disease course, barrier gestures, social distancing.
  Groups: Children
Other: Phone call interview — less than 15 minutes phone call
  Groups: Adults

SUMMARY:
Unlike other respiratory viruses such as influenza and RSV where the child is the essential reservoir and central vector of intrafamilial contamination, the child is likely to be a small player in the transmission of CoV2-CoRSA infection. This study aims to describe the age category of the first contact, within 14 days before the appearance of the first symptoms of the index case in order to describe the age categories of this first contaminant, globally, in the group of children and finally in the group of adults. This work is intended to provide food for discussion and to justify the distancing and containment measures imposed on children when their isolation has a deleterious impact that has now been established for some children.

ELIGIBILITY:
Inclusion Criteria:

* 1) Children hospitalized in the Pediatric department of the Hospices Civils de Lyon with PCR positive for a variant of the historical SARS-CoV2, 2) Adults hospitalized in the the Hospices Civils de Lyon, for a Covid-19 disease with documented infection by a variant of the SARS-CoV-2 and included in the NOSO-COR study with matching criteria described below.

Exclusion Criteria:

1. Any patient suspected of nosocomial infection.
2. Any patient death during the Covid-19 infection.
3. Any adult patient without children living home.
4. Opposition to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital-based population of children and adults:
  * Hospitalized children, 0 to 17 years of age, 25 subjects, consecutive sample survey
  * Hospitalized adults, 18 years and above, 50 matched subjects
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Percentage of possible contaminants, adults, adolescents and children with Covid-19 | At inclusion
  To describe the age category of the 1st possible contaminant in the index case to show the preponderance of possible adult and adolescent contaminants in the SARS-Cov-2 contamination.
  Primary endpoint: Percentage of possible contaminants, adults, adolescents and children, in matched children and adults with Covid-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère et enfant, Lyon, Auvergne-Rhône-Alpes, France